CLINICAL TRIAL: NCT05592483
Title: A Multi-center, Multi-country Prospective Observational Study of Patients Initiating T-DXd in the First or Second Treatment Line for HER2+, and HER2-low Unresectable and/or Metastatic Breast Cancer
Brief Title: An Observational Study of Patients Receiving T-DXd for Treatment of HER2+, and HER2-low Unresectable and/or Metastatic Breast Cancer
Acronym: DB RESPOND
Status: Terminated | Type: Observational
Why Stopped: The DESTINY-Breast RESPOND study was terminated early due to start-up delays and slow enrolment, despite extensive mitigation. Operational challenges alone prevent study continuation and were not related to any product or patient safety concerns.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9673R00025
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: Real-World Evidence; Unresectable Breast Cancer; Metastatic Breast Cancer; HER2+; HER2-low; Observational; non-interventional
MeSH Terms: conditions — Breast Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HER2+ Cohort: Patients with HER2+ unresectable and/or mBC who are prescribed T-DXd and have received a prior anti-HER2 based regimen.
  Interventions: Other: None (Observational Study)
- HER2-low cohort: Patients with HER2-low unresectable and/or mBC who are prescribed T-DXd and have received a prior chemotherapy.
  Interventions: Other: None (Observational Study)

INTERVENTIONS:
Other: None (Observational Study) — Not Applicable since observational study
  Other Names: Observational study

SUMMARY:
This study will collect real-world clinical and patient reported outcomes (PRO) and diary data from eligible patients with documented Human Epidermal Growth Factor Receptor 2 (HER2+) [globally] or HER2-low [North America only] in routine clinical practice.

DETAILED DESCRIPTION:
This is a multi-center, observational prospective study that will characterize the demographic and clinical characteristics, treatment patterns, effectiveness, tolerability and its management, and patient experience of Trastuzumab Deruxtecan (T-DXd) in a real-world setting. This study is planned to be conducted in several countries and aims to enroll approximately 750 patients eligible patients with HER2+ unresectable and/or metastatic breast cancer (mBC) who has received a prior anti HER2 based regimen in the metastatic setting or in the neoadjuvant or adjuvant setting and has developed disease recurrence during or within 6 months of completing therapy. Approximately 250 eligible patients with HER2-low unresectable and/or mBC who have received a prior chemotherapy in the metastatic setting or developed disease recurrence during or within 6 months of completing adjuvant chemotherapy will be enrolled into the study in North America only.

The planned duration of patient recruitment is approximately 18 months for HER2+ and approximately 12 months for HER2 low.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age at time of consent.
* Histological or cytological confirmed diagnosis of unresectable and/or mBC.
* Documented HER2 status via a validated method.
* Adult patients with unresectable or metastatic HER2+ breast cancer who have received a prior anti-HER2-based regimen in the metastatic setting or in the neoadjuvant or adjuvant setting and developed disease recurrence during or within 6 months of completing therapy.

Or

Adult patients with unresectable or metastatic HER2 low (IHC 1+ or IHC 2+/ISH-) breast cancer who have received a prior chemotherapy in the metastatic setting or developed disease recurrence during or within 6 months of completing adjuvant chemotherapy.

* Decision to newly initiate monotherapy T-DXd per standard of care.
* Capable of providing informed consent and completing questionnaires.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* History of other primary malignancies in 2 years prior to unresectable and/or mBC diagnosis.
* Patients who at time of data collection for this study are participating in or have participated in an interventional study that remains blinded.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HER2+ and HER2-low unresectable and/or mBC who are prescribed T-DXd for 2L or earlier metastatic treatment per standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Real-World Time to Next Treatment (rwTTNT) | From first dose of T-DXd until study discontinuation (approximately 3 years)
  Real-world time to next treatment will be evaluated. rwTTNT is defined as the length of time from date of first T-Dxd administration to the date the patient received an administration of their next systemic treatment regimen or to their date of death if there is a death prior to having another systemic treatment regimen.
T-Dxd treatment patterns for HER2+ cohort | Approximately 3 years
  Treatment patterns will be summarised using summary statistics.

SECONDARY OUTCOMES:
T-Dxd treatment patterns for HER2-low | Approximately 3 years
  Treatment patterns will be summarised using summary statistics.
Demographics and clinical charcteristics | At Baseline (14 to 30 days prior to T-DXd initiation)
  Summary statistics will be used to describe the Demographics and clinical characteristics
Number of patients with Physician reported Safety Events of Interest (SEIs) | From first dose of T-DXd until End of T-DXd treatment (40 + 7 days after last T-DXd administration)
  The safety and tolerability of T-Dxd through the collection of physician-reported SEIs will be assessed.
Number of patients provided prophylactic and reactive treatment for SEIs management | From first dose of T-DXd until End of T-DXd treatment (40 + 7 days after last T-DXd administration)
  The management of SEIs will be characterized.
Real-World Time to Discontinuation (rwTTD) | From first dose of T-DXd until study discontinuation (approximately 3 years)
  Real-World Time to Discontinuation of T-DXd will be evaluated. rwTTD is defined as time from index date to the earliest date of T-DXd discontinuation, or death.
Patient-reported overall side effect burden as measured by the Patient's Global Impression of Treatment Tolerability (PGI-TT) | Approximately 3 years
  Patient-reported tolerability will be evaluated by PGI-TT. Single question asking patients how bothered they were by the side effects of their cancer treatment, ranging from Not at all to Very much.
Symptomatic SEI as measured by selected items from National Cancer Institute Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (NCI PRO-CTCAE) | Approximately 3 years
  Patient-reported tolerability will be evaluated by selected items from the NCI PRO-CTCAE. The following items are selected: nausea, vomiting, bloating of the abdomen, shortness of breath, cough, heart palpitations, hair loss, and fatigue, tiredness or lack of energy.
Daily Nausea and Vomiting symptom diary | From first dose of T-DXd until 3 months
  Nausea and vomiting symptoms diary will be assessed based on severity, interference with appetite and usual activities.

CONTACTS AND LOCATIONS:
Locations (117):
- United States (39):
  - Research Site, Mobile, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Los Angeles, California
  - Research Site, Santa Rosa, California
  - Research Site, Pensacola, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Evergreen Park, Illinois
  - Research Site, Glenview, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Annapolis, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Southfield, Michigan
  - Research Site, Saint Paul, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, Camden, New Jersey
  - Research Site, Florham Park, New Jersey
  - Research Site, Jamaica, New York
  - Research Site, Lake Success, New York
  - Research Site, Eugene, Oregon
  - Research Site, York, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Germantown, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, McAllen, Texas
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tyler, Texas
  - Research Site, Portsmouth, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Everett, Washington
  - Research Site, Milwaukee, Wisconsin
- Austria (5):
  - Research Site, Vienna, Nordrhein-Westfalen
  - Research Site, Graz, Styria
  - Research Site, Innsbruck, Tyrol
  - Research Site, Wels, Upper Austria
  - Research Site, Vienna
- Brazil (9):
  - Research Site, Cachoeiro de Itapemirim, Espírito Santo
  - Research Site, Salvador, Estado de Bahia
  - Research Site, Brasília, Federal District
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Curitiba, Paran
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Itajaí
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Canada (7):
  - Research Site, Calgary, Alberta
  - Research Site, Surrey, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Kingston, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec
- Israel (4):
  - Research Site, Jerusalem, Jerusalem
  - Research Site, Tel Aviv, Tel Aviv
  - Research Site, Beersheba
  - Research Site, Haifa
- Italy (9):
  - Research Site, Brescia
  - Research Site, Brindisi
  - Research Site, Catania
  - Research Site, Cremona
  - Research Site, Palermo
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Torino
  - Research Site, Verona
- Spain (31):
  - Research Site, A Coruña, A Coruna
  - Research Site, Elche, Alicante
  - Research Site, Zaragoza, Aragon
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, L'Hospitalet de Llobregat, Barcelona
  - Research Site, Jerez de la Frontera, Cadiz
  - Research Site, Las Palmas de Gran Canaria, Canary Islands
  - Research Site, Santa Cruz de Tenerife, Canary Islands
  - Research Site, Santander, Cantabria
  - Research Site, Ourense, Galicia
  - Research Site, Donostia / San Sebastian, Guipuzcoa
  - Research Site, Logroño, La Rioja
  - Research Site, Madrid, Madrid
  - Research Site, Majadahonda, Madrid
  - Research Site, Pamplona, Navarre
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Reus, Tarragona
  - Research Site, Barakaldo, Vizcaya
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Cáceres
  - Research Site, Córdoba
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Segovia
  - Research Site, Seville
  - Research Site, Toledo
  - Research Site, Valencia
  - Research Site, Zaragoza
- Switzerland (4):
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Liestal
  - Research Site, Monthey
- United Kingdom (9):
  - Research Site, Keighley, England
  - Research Site, Rickmansworth, England
  - Research Site, Londonderry, Northern Ireland
  - Research Site, Inverness, Scotland
  - Research Site, Taunton, Somerset
  - Research Site, Coventry
  - Research Site, Huddersfield
  - Research Site, Leeds
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR not created for the study-rationale — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9673R00025&attachmentIdentifier=d4d4254c-5414-40a6-9425-a1932c7ac28d&fileName=D9673R00025_Statement.pdf&versionIdentifier=